CLINICAL TRIAL: NCT02080923
Title: A Brief Intervention to Prevent Adolescent Dating Aggression Perpetration
Acronym: PLR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-31501; 2013-VA-CX-0001 (Other Grant/Funding Number: Sponsor Name: National Institute of Justice)
Record Dates: First submitted 2014-03-04; First posted 2014-03-07 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-06

CONDITIONS: Offensive Aggression; Sexual Aggression; Dating Violence Perpetration and Victimization
Keywords: Adolescent; Adolescent Behavior; Age Factors; Courtship; Randomized Control Trial; Female; Male; Minority Groups/statistics & numerical data; Risk-Taking; Sex Factors; Sexual Behavior/statistics & numerical data; Substance-Related Disorders/epidemiology; Urban Population/statistics & numerical data; Violence/statistics & numerical data; Dating Violence; Dating Aggression; Perpetration
MeSH Terms: conditions — Adolescent Behavior; Courtship; Risk-Taking; Sexual Behavior; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: This is a brief motivational interview-style intervention. Adolescents ages 15-19 years old who visit the emergency department and screen positive for physical or sexual dating abuse perpetration participate in a ~45 minute brief intervention and receive up to three booster calls in the subsequent 6 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Motivational Interview (Experimental): Health-related counseling that takes place in as little as one hour or up to a few sessions.
  Interventions: Behavioral: Brief Motivational Interview
- Standard Care (No Intervention): Participant will receive information about dating abuse in a handout and referrals to a national domestic violence hotline.

INTERVENTIONS:
Behavioral: Brief Motivational Interview — The intervention is exclusively focused on Adolescent Dating Aggression and will always be delivered by a human interventionist. It is theory-based and its success as an intervention method for substance abuse and several other health-related issues is well established.
  Arms: Brief Motivational Interview

SUMMARY:
The proposed study is a test of the feasibility and preliminary efficacy of a brief motivational interview style intervention. The intervention will take place in the pediatric emergency department of the Boston University Medical Center by a trained interventionist and will follow an intervention manual developed by a team of dating abuse and brief intervention experts. The study will involve two randomized groups of youth age 15-19: one group will receive the intervention and the other will not. The study will compare changes in data from baseline to 3- and 6-month follow-up for those in both groups. Outcomes including dating abused related knowledge, attitudes about the use of violence to resolve conflict, and dating abuse behavior (perpetration and/or victimization) will be assessed.

The hypothesis of this study is that youth who receive the intervention will show improvements in dating abuse related knowledge, attitudes and behavior that are maintained for 6 months, while those in the control group will show no similar change.

DETAILED DESCRIPTION:
Emergency departments offer a unique setting through which we can reach adolescents who have perpetrated Adolescent Dating Aggression (ADA). The Project READY (Reducing Aggression in Dating Relationships for Youth) brief intervention manual and training was developed by Dr. Emily Rothman, who is a former shelter worker, batterer intervention counselor, and dating violence expert, with input from research experts in brief intervention, an expert in adolescent batterer intervention, psychologists, low-income youth of color from the Start Strong Initiative, and others, with funding from the National Institutes of Health (NIH). The READY intervention intercepts youth who utilize an urban emergency department for non-acute health care needs (e.g., cuts, sprains), provides them with tailored feedback about their relationship behavior, and uses motivational interviewing techniques and prepared worksheets to move them forward on a readiness-to-change continuum towards non-violent and respectful relationship behavior. For example, after being provided with information about acts considered unhealthy in a relationship, a participant is asked to generate a list of "pros and cons" about what he or she does to solve conflicts with partners, brainstorm alternatives that he or she would use, list reasons why the alternatives might not work in the moment, and troubleshoot those potential problems. Participants are then offered a menu of referrals and invited to select those that they would use (e.g., free mental health and substance abuse counseling, sexual health testing, gang prevention resources).

The randomized controlled trial (RCT) research study will build upon our completed small-scale feasibility pilot project, which was conducted in 2012- 13. For the proposed study, we will recruit a sample large enough to evaluate whether the intervention improves ADA-related knowledge, positively changes ADA-related attitudes and behavioral intentions, and reduces self-reported perpetration behavior after 3- and 6-month follow-up periods. The study will enroll youth ages 15-19 years old. Notably, the setting for this intervention test will be an urban pediatric emergency department that primarily serves low income youth.

ELIGIBILITY:
Inclusion Criteria:

* must be a patient of the Pediatric Emergency Department or adolescent outpatient center at the Boston University Medical Center
* must be 15-19 years old
* have used at least one form of physical or sexual aggression against a dating or sexual partner in the past three months
* English-speaking

Exclusion Criteria:

* patient's reason for visit to the healthcare center is an acute mental health problem
* patient is a prisoner or juvenile detainee
* patient is determined to be a potentially lethal dating abuse offender based on a lethality checklist
* patient has cognitive or psychiatric limitations that render him/her unable to complete the eligibility form independently
* currently attending a batterer intervention program
* receiving care for violent trauma victimization
* appears intoxicated or high on drugs at the time of eligibility screening, or has informed medical staff that they are

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 220 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
Dating Aggression Perpetration | 3 months or 6 months
  Change in the perpetration of dating aggression from baseline to follow-up.
Intentions to use physical violence during next partner conflict | 3 months or 6 months
  Change in the intention to use acts of physical violence during the next conflict with a dating partner

SECONDARY OUTCOMES:
Knowledge and Attitudes about Dating Aggression | 3 months or 6 months
  Change in Knowledge and Attitudes about Dating Aggression from baseline to the three month follow-up

OTHER OUTCOMES:
Program Cost-effectiveness | up to 18 months
  Costs are the value of resources used before and during implementation to deliver the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Emily F Rothman, MS, ScD, Principal Investigator — Boston University
Locations (1):
- Boston University School of Public Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rothman EF, Stuart GL, Heeren T, Paruk J, Bair-Merritt M. The Effects of a Health Care-Based Brief Intervention on Dating Abuse Perpetration: Results of a Randomized Controlled Trial. Prev Sci. 2020 Apr;21(3):366-376. doi: 10.1007/s11121-019-01054-w. PMID 31643025
- See also: Academic Profile — http://profiles.bu.edu/Emily.Rothman